CLINICAL TRIAL: NCT00936884
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, And Parallel-Group Study Of Subcutaneous Methylnaltrexone (MOA-728) For The Treatment Of Opioid-Induced Constipation In Adult Subjects
Brief Title: Study Evaluating the Efficacy and Safety of Subcutaneous Methylnaltrexone (MOA-728) for the Treatment of Opioid-Induced-Constipation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Collaborators: Progenics Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3200K1-3361; B2541004
Record Dates: First submitted 2009-07-08; First posted 2009-07-10 (Estimated); Results first posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Constipation
Keywords: Opioid Induced Constipation
MeSH Terms: conditions — Constipation; Opioid-Induced Constipation | interventions — methylnaltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Methylnaltrexone double-blind (Experimental): Methylnaltrexone once every other day.
  Interventions: Drug: Methylnaltrexone
- Placebo (Placebo Comparator): Placebo once every other day.
  Interventions: Drug: Placebo
- Methylnaltrexone open-label (Other): Subjects who completed the double-blind period had the option to receive methylnaltrexone once every other day during a 12-week, open-label extension period.
  Interventions: Drug: Methylnaltrexone

INTERVENTIONS:
Drug: Methylnaltrexone — Subjects received 0.6 mL (12 mg) every other day if weight ≥ 62kg; 0.4 mL (8 mg) every other day if weight between 38 and < 62 kg; or 0.0075 mL/kg (0.15 mg/kg) every other day if weight between 27 and <38 kg.
  Study duration: 2 weeks double-blind period (MNTX treatments) followed by 12 weeks open-label extension period (MNTX treatments).
  Other Names: MOA-728; MNTX
  Arms: Methylnaltrexone double-blind; Methylnaltrexone open-label
Drug: Placebo — Subjects received matching placebo injections.
  Study duration: 2 weeks double-blind period (placebo treatments) followed by 12 weeks open-label extension period (MNTX treatments).
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to evaluate the safety, efficacy, and tolerability of subcutaneous (injection beneath the skin) MOA-728 versus placebo in adult Asian subjects with opioid-induced constipation associated with advanced illness (ie, a terminal illness such as incurable cancer or other end-stage disease) or chronic nonmalignant pain.

DETAILED DESCRIPTION:
Subjects received subcutaneous methylnaltrexone (also referred to as MOA-728 or MNTX) or placebo every other day beginning on Day 1 up to a maximum of 7 doses during the 2-week double-blind period.

Inclusion criteria for this study included subjects with advanced illness or subjects with chronic nonmalignant pain. The actual study population included only subjects with cancer-related advanced illness.

All subjects who completed the double-blind treatment phase of this study could elect to receive methylnaltrexone during a 12-week open-label extension study, provided eligibility criteria were met. Subjects who did not continue in the open-label extension study had a follow-up visit 2 weeks after their last dose of test article.

ELIGIBILITY:
Inclusion Criteria:

* Men and women who are at least 18 years of age, and who have a diagnosis of advanced illness with anticipated life expectancy >= 1 month;
* Is receiving a regular dose of opioids for the control of pain;
* Has a diagnosis of opioid induced constipation;
* Is on a stable laxative regimen.

Exclusion Criteria:

* Has a known or suspected mechanical gastrointestinal obstruction, or any potential non-opioid cause of bowel dysfunction contributed to constipation;
* Has evidence of current fecal impaction;
* Has evidence of active diverticulitis, or peritonitis, or a history of bowel surgery within 30 days before test article administration;
* Has a body weight less than 27 kg
* Has any major illness/condition that, in the investigator's judgment, will substantially increase the risk associated with the subject's participation in and completion of the study, or could preclude the evaluation of the subject's response.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-07; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Enoch Bortey, Study Director — Bausch Health Americas, Inc.
Locations (4):
- South Korea (2):
  - Koyang-shi, Kyounggi-do
  - Seoul
- Taiwan (2):
  - Tainan
  - Taipei TOC

RESULTS

PARTICIPANT FLOW:
Period: Double-blind
Arm/Group | Methylnaltrexone Double-blind | Placebo | Methylnaltrexone Open-label
Started | 25 (Twenty-five subjects received MNTX, and 24 had ≥ 1 post baseline diary assessment.) | 25 (Twenty-four subjects received placebo, and 23 had ≥ 1 post baseline diary assessment.) | 0 (Thirteen subjects from the MNTX group and 18 from the placebo group entered the 12-week extension.)
Completed | 13 | 18 | 0
Not Completed | 12 | 7 | 0
Not completed — Withdrawal by Subject | 6 | 4 | 0
Not completed — Death | 2 | 1 | 0
Not completed — Lack of Efficacy | 1 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — No post baseline diary entry | 1 | 0 | 0
Not completed — Did not receive study drug | 0 | 1 | 0
Period: Open-label
Arm/Group | Methylnaltrexone Double-blind | Placebo | Methylnaltrexone Open-label
Started (Thirteen subjects from the MNTX group and 18 from the placebo group entered the 12-week extension.) | 0 | 0 | 31
Completed | 0 | 0 | 12
Not Completed | 0 | 0 | 19

BASELINE CHARACTERISTICS:
Population: All randomized subjects were included in the baseline population. Patients in the MNTX open-label group included subjects who had already participated in the MNTX double-blind or placebo groups during the double-blind period. Therefore, baseline characteristics are not repeated for the subjects who continued in the open-label extension period.
Groups:
- Methylnaltrexone Double-blind: Methylnaltrexone once every other day.
  Subjects received 0.6 mL (12 mg) every other day if weight ≥ 62kg; 0.4 mL (8 mg) every other day if weight between 38 and < 62 kg; or 0.0075 mL/kg (0.15 mg/kg) every other day if weight between 27 and <38 kg.
- Placebo: Placebo once every other day.
  Subjects received matching placebo injections.
- Total: Total of all reporting groups
Arm/Group | Methylnaltrexone Double-blind | Placebo | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 13 | 31
  >=65 years | 7 | 12 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (11.68) | 62.1 (14.23) | 60.3 (13.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 11 | 25
  Male | 11 | 14 | 25
Eastern Cooperative Oncology Group Score [Count of Participants; unit: Participants]
  0 - Fully active | 0 | 1 | 1
  1 - Restricted in strenuous activity | 3 | 4 | 7
  2 - Unable to work | 6 | 5 | 11
  3 - Limited self-care | 16 | 15 | 31
Hospitalization Status at Screening Period [Number; unit: participants]
  Yes | 12 | 8 | 20
  No | 13 | 17 | 30
Underlying Advanced Illness - Cancer-related illness [Count of Participants; unit: Participants] | 25 | 25 | 50
Weight [Count of Participants; unit: Participants]
  < 38 kg | 2 | 0 | 2
  38 - < 62 kg | 17 | 20 | 37
  ≥62 kg | 6 | 4 | 10
  Missing | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Subjects Having a Rescue-free Bowel Movement (RFBM) Within 4 Hours After the First Injection.
Description: There were 2 co-primary endpoints for this study. This measurement is the first of the 2 co-primary endpoints. This endpoint measures the percentage of patients who had an RFBM within 4 hours after the first dose of test article during the double-blind period; data are expressed as percentages of patients for the MNTX and placebo groups. To qualify as rescue free, the bowel movement could not occur within 6 hours after a rectal intervention (ie, rectal suppository, enema, manual disimpaction). Note that efficacy results (primary and secondary outcomes) are presented for the double-blind period only. Therefore, no efficacy results are presented for the open-label period.
Time Frame: Up to 4 hours after the first injection
Population: Although 25 patients in the MNTX group and 24 in the placebo group received study drug, 24 and 23 patients, respectively, had ≥ 1 post baseline diary assessment and were analyzed for efficacy.
Measure: Number; unit: percentage of participants
Arm/Group | Methylnaltrexone Double-blind | Placebo
Number analyzed (Participants) | 24 | 23
percentage of participants | 79.2 | 4.3
Statistical Analysis 1: Comparison: Methylnaltrexone Double-blind vs Placebo; Test type: Superiority or Other; p < 0.0001, Chi-squared — Comparison of the MNTX group and the placebo group in the proportion of subjects having a RFBM within 4 hours after the first injection was performed by using a 2-sided Cochran-Mantel-Haenszel Chi square test at the alpha level of 0.025; Odds Ratio (OR) = 83.60, 97.5% CI 2-sided [6.50 to 1074.7]

2. Secondary Outcome: Percentage of Injections Resulting in RFBM Within 4 Hours After Test Article Administration.
Description: This endpoint measures the percentage of injections resulting in RFBMs within 4 hours after test article administration during the double-blind period. The percentage of injections resulting in RFBMs is calculated for each patient and then data are expressed as the mean (± standard deviation) percentage for the MNTX and placebo groups. The definition of RFBM is described above (see first co-primary endpoint).
Time Frame: Within 4 Hours After Each Dose During the 2 weeks Double-Blind Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of injections
Arm/Group | Methylnaltrexone Double-blind | Placebo
Number analyzed (Participants) | 24 | 23
percentage of injections | 61.61 (36.520) | 4.97 (22.203)
Statistical Analysis 1: Comparison: Methylnaltrexone Double-blind vs Placebo; Test type: Superiority or Other; p < 0.0001, ANOVA — Comparison of the MNTX group and the placebo group was based on ANOVA model with the proportion of injections resulting in RFBM within 4 hours during the double-blind period as the dependent variable and the treatment group as the fixed effect; Mean Difference (Final Values) = 56.64, 97.5% CI 2-sided [40.62 to 72.66] — Estimated value is the difference in least squared means for MNTX vs. placebo (MNTX minus placebo). Based on the ANOVA model, there is 97.5% confidence that the difference between MNTX and placebo falls between the lower and upper limits presented

3. Primary Outcome: The Proportion of Subjects Having a Rescue-free Bowel Movement (RFBM) Within 4 Hours After Each Dose During Double-blind Period.
Description: This measurement is the second of the 2 co-primary endpoints. This endpoint measures the percentage of patients who had an RFBM within 4 hours after each dose of test article during the double-blind period; data are expressed as percentages of patients by dose (first, second, third, fourth, etc.) for the MNTX and placebo groups. The definition of RFBM is described above (see first co-primary endpoint).
Time Frame: Within 4 Hours After Each Dose During the 2 weeks Double-Blind Period
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Methylnaltrexone Double-blind | Placebo
Number analyzed (Participants) | 24 | 23
percentage of participants
  RFBM post second DB injection | 61.9 | 8.7
  RFBM post third DB injection | 52.6 | 8.7
  RFBM post fourth DB injection | 38.9 | 8.7
  RFBM post fifth DB injection | 56.3 | 4.5
  RFBM post sixth DB injection | 43.8 | 0
  RFBM post seventh DB injection | 43.8 | 0
  RFBM post eighth DB injection | 57.1 | 7.7
Statistical Analysis 1: Comparison: Methylnaltrexone Double-blind vs Placebo; Test type: Superiority or Other; p < 0.0001, Chi-squared — Comparison of the MNTX group and the placebo group in the proportion of subjects having a RFBM within 4 hours after each injection was performed by using a 2-sided Cochran-Mantel-Haenszel Chi square test at the alpha level of 0.025; Odds Ratio (OR) = 23.38, 97.5% CI 2-sided [10.91 to 50.14]

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the 2-week double-blind period and over the 12-week open-label period.
Description: Adverse events were collected by non-systematic (patient reports) and systematic methods (investigator examinations and lab tests). For both adverse events tables, a subject reporting more than one adverse event for a particular MedDRA preferred term or system organ class was counted only once for that MedDRA preferred term or system organ class.
Arm/Group | Methylnaltrexone Double-blind | Placebo | Methylnaltrexone Open-label
Serious Adverse Events (participants affected / at risk) | 12/25 | 8/24 | 21/31
Other Adverse Events (participants affected / at risk) | 16/25 | 18/24 | 25/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Methylnaltrexone Double-blind (N=25) | Placebo (N=24) | Methylnaltrexone Open-label (N=31)
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 2
Nausea (Gastrointestinal disorders) | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
Asthenia (General disorders) | 1 | 2 | 9
Disease progression (General disorders) | 0 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 4
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 5 | 9
Somnolence (Nervous system disorders) | 1 | 0 | 2
Dysuria (Renal and urinary disorders) | 0 | 1 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Malignant neoplasm progression (General disorders) | 0 | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Chest discomfort (General disorders) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Mesothelioma malignant advanced (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Diplegia (Nervous system disorders) | 1 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 1
Melena (Gastrointestinal disorders) | 0 | 0 | 1
Feeling cold (General disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Methylnaltrexone Double-blind (N=25) | Placebo (N=24) | Methylnaltrexone Open-label (N=31)
Anemia (Blood and lymphatic system disorders) | 1 | 3 | 4
Abdominal distension (Gastrointestinal disorders) | 2 | 2 | 3
Abdominal pain (Gastrointestinal disorders) | 4 | 1 | 2
Ascites (Gastrointestinal disorders) | 4 | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 4
Nausea (Gastrointestinal disorders) | 1 | 2 | 2
Vomiting (Gastrointestinal disorders) | 2 | 1 | 3
Asthenia (General disorders) | 0 | 1 | 9
Edema (General disorders) | 0 | 1 | 3
Edema peripheral (General disorders) | 3 | 0 | 3
Fatigue (General disorders) | 0 | 2 | 0
Pain (General disorders) | 2 | 0 | 1
Pyrexia (General disorders) | 3 | 1 | 1
Jaundice (Hepatobiliary disorders) | 1 | 2 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1 | 7
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3
Dizziness (Nervous system disorders) | 3 | 1 | 1
Headache (Nervous system disorders) | 0 | 1 | 2
Somnolence (Nervous system disorders) | 2 | 1 | 2
Dysuria (Renal and urinary disorders) | 4 | 3 | 1
Delirium (Psychiatric disorders) | 1 | 0 | 2
Insomnia (Psychiatric disorders) | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 0 | 1
Hypotension (Vascular disorders) | 1 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less